CLINICAL TRIAL: NCT05213208
Title: Propofol Sedation of More Than 200 mg Enables Patients to Drive Home After Outpatient Colonoscopy Including Colorectal Polypectomy
Brief Title: Safety of Propofol Sedation ( > 200 mg) for Colonoscopy.
Status: Completed | Type: Observational
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Other Study IDs: PS>200
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Safety Issues
Keywords: driving; propofol sedation; colonoscopy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Propofol — Using > 200 mg of propofol sedation colonoscopy is performed. 90-120 minutes after colonoscopy subjects go home. Within 1 week patients will be asked about their condition and satisfaction for colonoscopy.

SUMMARY:
This study examines that the use of >200 mg of propofol sedation enables patients to drive home safely after outpatient colonoscopy.

DETAILED DESCRIPTION:
The hospital policy of routine discharge to normal activity 1 hour after propofol mono-sedation for EGD or colonoscopy was approved by the ethics committee of Showa Inan General Hospital in January, 2004 (http://www.sihp.jp). The investigator' s subsequent experience verified the safety of this discharge policy which was reconfirmed in March 2014. Based on these studies, the upper limit of 200 mg was established for those allowed early discharge and driving to home.

This study examines that the use of >200 mg of propofol sedation enables patients to drive home safely 90-120 minutes after outpatient colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* subjects who drive home by theirselves after colonoscopy using propofol sedation (>200 mg)

Exclusion Criteria:

* Subjects who received emergency procedures
* less than 20 years old pregnant American Society of Anesthesiologists (ASA) class III or IV, overweight (body weight >100 kg) allergic to the drugs used or its components (soybeans or eggs).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: healthy subjects who drive home after colonoscopy using propofol sedation (>200 mg)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Traffic accidents | 1 day
  Number of traffic accidents

SECONDARY OUTCOMES:
Patient satisfaction | 1 day
  Patient satisfaction (bad, 0-good 100%) is asked.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horiuchi I, Horiuchi K, Kitahara H, Horiuchi A. Does >200 mg of Propofol Sedation Allow Healthy Individuals to Undergo a Colonoscopy and Drive Themselves Home? J Clin Gastroenterol. 2025 Sep 30. doi: 10.1097/MCG.0000000000002252. Online ahead of print. PMID 41071172